CLINICAL TRIAL: NCT00386477
Title: Vaginal Cleansing at Cesarean Delivery to Reduce Infection: A Randomized, Controlled Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty recruiting
Sponsor: Indiana University School of Medicine (Other)
Responsible Party: David M. Haas/ Assistant Professor of OB/GYN, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0509-55 (Study #); 0509-55 (Other: IUPUI-Clarian IRB number)
Record Dates: First submitted 2006-10-09; First posted 2006-10-11 (Estimated); Results first posted 2010-02-08 (Estimated); Last update posted 2010-02-08 (Estimated); Status verified 2010-12

CONDITIONS: Cesarean Section; Endometritis; Surgical Wound Infection
Keywords: Povidone iodine; postoperative infection; presurgical cleansing
MeSH Terms: conditions — Endometritis; Surgical Wound Infection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vag prep (Experimental): Vagina cleansed prior to performing cesarean
  Interventions: Procedure: Vaginal cleansing before cesarean delivery

INTERVENTIONS:
Procedure: Vaginal cleansing before cesarean delivery — Cleansing vagina with 1% betadine scrub before cesarean.
  Other Names: 1% betadine scrub of vagina with vaginal scrub spongesticks.

SUMMARY:
The objective of the project is to find out whether cleansing the vagina before a cesarean delivery decreases the risk of complications and infections after having the baby. If this is the case, cleansing the vagina before cesarean delivery can help improve outcomes for many women and make their early postpartum recovery much more pleasant, giving a healthier start for the family.

DETAILED DESCRIPTION:
Infectious morbidity frequently complicates cesarean delivery. Endometritis can complicate the postoperative course of a cesarean delivery 6-27% of the time. This complication, up to 10 times more frequent than after vaginal delivery, can lead to serious complications. Additionally, cesarean deliveries are frequently complicated by maternal fever and wound complications including seroma, hematoma, infection, and separation. These morbidities can lead to significant delay in a return to normal function. Our study will randomize 1000 women who are about to undergo a cesarean delivery into one of two groups. The control group will receive the standard surgical preparation of the abdomen alone, the current standard pre-cesarean preparation. The other group will also receive a povidone iodine washing/scrub of the vagina before the cesarean delivery. Maternal and surgical variables will be recorded. At one months postpartum, maternal outpatient data will be reviewed and the incidence of postpartum uterine infection, wound separations, and other wound and infectious complications will be determined and compared between the two treatment groups.

Comparison: Women receiving standard surgical abdominal cleansing versus women receiving standard abdominal and preoperative vaginal cleansing before cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* Woman undergoing cesarean delivery
* At least 18 years of age

Exclusion Criteria:

* Allergy to iodine containing solutions
* Planned cesarean hysterectomy
* Prisoner

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2006-09; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Haas, MD, Principal Investigator — Indiana University School of Medicine
Locations (3):
- United States (3):
  - Methodist Hospital, Indianapolis, Indiana
  - University Hospital, Indianapolis, Indiana
  - Wishard Memorial Hospital, Indianapolis, Indiana

REFERENCES:
- [Derived] Haas DM, Morgan S, Contreras K, Kimball S. Vaginal preparation with antiseptic solution before cesarean section for preventing postoperative infections. Cochrane Database Syst Rev. 2020 Apr 26;4(4):CD007892. doi: 10.1002/14651858.CD007892.pub7. PMID 32335895
- [Derived] Haas DM, Pazouki F, Smith RR, Fry AM, Podzielinski I, Al-Darei SM, Golichowski AM. Vaginal cleansing before cesarean delivery to reduce postoperative infectious morbidity: a randomized, controlled trial. Am J Obstet Gynecol. 2010 Mar;202(3):310.e1-6. doi: 10.1016/j.ajog.2010.01.005. PMID 20207251

RESULTS

PARTICIPANT FLOW:
Groups:
- Vag Prep: Vagina cleansed with betadine vaginal scrub sticks prior to performing cesarean
- Control: No vaginal cleansing or sham wash performed.
Period: Overall Study
Arm/Group | Vag Prep | Control
Started | 155 | 145
Completed | 155 | 145
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vag Prep | Control | Total
Number analyzed (Participants) | 155 | 145 | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 155 | 145 | 300
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 26.8 (5.9) | 26.6 (5.7) | 26.7 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 155 | 145 | 300
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants] — African-American Caucasian Hispanic Other
  participants | 155 | 145 | 300
Region of Enrollment [Number; unit: participants]
  United States | 155 | 145 | 300

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Composite Endometritis Plus Wound Complications.
Description: Endometritis was diagnosed clinically as uterine pain and fever requireing antibiotics. Wound complications included wound infection, seroma, hematoma, or separation.
Time Frame: 1 month
Population: Randomization
Measure: Number; unit: participants
Arm/Group | Vag Prep | Control
Number analyzed (Participants) | 155 | 145
participants | 10 | 17
Statistical Analysis 1: Comparison: Vag Prep vs Control; Test type: Superiority or Other; p = 0.11, Chi-squared, Corrected; Risk Ratio (RR) = 0.55, 95% CI [0.26 to 1.11]

ADVERSE EVENTS:
Time Frame: Adverse events would include any allergic or other reaction to the iodine vaginal cleansing.
Arm/Group | Vag Prep | Control
Serious Adverse Events (participants affected / at risk) | 0/155 | 0/145
Other Adverse Events (participants affected / at risk) | 0/155 | 0/145

LIMITATIONS AND CAVEATS:
The study was stopped before the planned enrollment of 1000 due to difficulty recruiting. Results are of a planned safety analysis at 300 subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No